CLINICAL TRIAL: NCT03468634
Title: Raman Probe for In-vivo Diagnostics (During Oesophageal) Endoscopy
Acronym: RaPIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: University of Bristol (Other); Gloucestershire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1516/017/162347; II-LB-0315-20008 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2018-01-11; First posted 2018-03-16 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Barrett Esophagus; Esophageal Cancer
Keywords: endoscopy; Raman spectroscopy
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms | interventions — Endoscopy; Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Adenocarcinoma (Experimental): patients diagnosed with adenocarcinoma
  Interventions: Diagnostic Test: endoscopy
- Squamous cell cancer (Experimental): patients diagnosed with squamous cell cancer
  Interventions: Diagnostic Test: endoscopy
- Other (Experimental): patients diagnosed with another condition
  Interventions: Diagnostic Test: endoscopy
- Barrett's oesophagus (Experimental): patients diagnosed with Barrett's oesophagus
  Interventions: Diagnostic Test: endoscopy
- Low-grade dysplasia (Experimental): patients diagnosed with low-grade dysplasia
  Interventions: Diagnostic Test: endoscopy
- High-grade dysplasia (Experimental): patients diagnosed with high-grade dysplasia
  Interventions: Diagnostic Test: endoscopy
- Indefinite for dysplasia (Experimental): patients where the diagnosis is unclear
  Interventions: Diagnostic Test: endoscopy
- no dysplasia (Experimental): patients not diagnosed with any cancer
  Interventions: Diagnostic Test: endoscopy

INTERVENTIONS:
Diagnostic Test: endoscopy — Oesophageal endoscopy with biopsy
  Other Names: EGD (esophagogastro duodenoscopy); upper GI endoscopy

SUMMARY:
To develop and endoscopic Raman spectroscopy probe for delivery down and channel in an endoscope to make near instant assessments of the condition of the oesophagus without the need for expensive and distressing tissue removal (biopsies).

DETAILED DESCRIPTION:
The investigators have already shown that it is possible to tell the difference between healthy and diseased tissue in the laboratory by looking at the light emitted by tissue when illuminated with a low power laser. The investigators intend to use this technique, known as "Raman Spectroscopy" to tell if tissue in the oesophagus is cancerous, healthy or at some stage before full blown cancer, which is termed pre-cancer. It has been shown in the laboratory that this method will be at least as accurate as the conventional methods used now, but will provide the surgeon with instant results without the delay and cost of a laboratory analysis by pathologists.

A miniature probe has been developed that slides through a channel in the endoscope (telescope) to the surface of the oesophagus to make near instant assessments of its condition without the need for expensive and distressing tissue removal (biopsies). This project plans to move this technique from the laboratory to the clinic by demonstrating that the method is safe and reliable for use in real patients.

ELIGIBILITY:
Inclusion Criteria:

* Barrett's oesophagus

Exclusion Criteria:

* Unfit for endoscopic and biopsy assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Device safety testing (no detectable damage in biopsy samples when reviewed by histopathology) | 6 months
  Testing of the device for clinical application to demonstrate its use is safe and that is able to acquire diagnostic-quality (see outcome 2) spectra in less than 5 seconds from within the oesophagus.
  Samples illuminated will be biopsied and sent for routine histopathological analysis.

SECONDARY OUTCOMES:
Diagnostic model developed (algorithm able to discriminate disease with >50% specificity and >50% sensitivity) | 6 months
  Computer model using multivariate analysis able to discriminate between diseased and non-diseased tissue. The target specificity and sensitivity are low due to small study group sizes.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Old, BMedSc MBChB, Principal Investigator — Gloucestershire Hospitals NHS Foundation Trust
Locations (1):
- Gloucestershire Hospitals NHS Foundation Trust, Gloucester, Gloucestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Isabelle M, Dorney J, Lewis A, Lloyd GR, Old O, Shepherd N, Rodriguez-Justo M, Barr H, Lau K, Bell I, Ohrel S, Thomas G, Stone N, Kendall C. Multi-centre Raman spectral mapping of oesophageal cancer tissues: a study to assess system transferability. Faraday Discuss. 2016 Jun 23;187:87-103. doi: 10.1039/c5fd00183h. PMID 27048868
- [Background] Kendall C, Stone N, Shepherd N, Geboes K, Warren B, Bennett R, Barr H. Raman spectroscopy, a potential tool for the objective identification and classification of neoplasia in Barrett's oesophagus. J Pathol. 2003 Aug;200(5):602-9. doi: 10.1002/path.1376. PMID 12898596
- See also: RaPIDE project website — https://rapide-diagnostics.co.uk/